CLINICAL TRIAL: NCT04003714
Title: EFFECTIVENESS OF REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION IN PATIENTS WITH FAILED BACK SURGERY SYNDROME A DOUBLE-BLINDED, RANDOMISED, PLACEBO CONTROLLED TRIAL
Brief Title: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION FOR FAILED BACK SURGERY SYNDROME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: meryemyılmazkaysın
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Failed Back Surgery Syndrome
Keywords: repetitive transcranial magnetic stimulation; back pain; failed back surgery syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome; Back Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive Transcranial Magnetic Stimulation Group (Experimental): Patients in r-TMS group received r-TMS 20-min (1000 pulses) daily session, 5 days per weeks, for a total of 10 sessions.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham Group (Sham Comparator): Control group received sham r-TMS with the same protocol.
  Interventions: Device: Sham Repetitive transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Patients in r-TMS group received 5 Hz of r-TMS. R-TMS applied with MagVenture device (MagPro X100, Denmark, 2009) and figure eight coil (MMC 140 parabolic, MagVenture).
  Arms: Repetitive Transcranial Magnetic Stimulation Group
Device: Sham Repetitive transcranial Magnetic Stimulation — Control group received sham r-TMS.
  Arms: Sham Group

SUMMARY:
Failed back surgery syndrome (FBSS) is the term of persistent back and/or leg pain after surgery for lumbar disk herniation (LDH). Repetitive transcranial magnetic stimulation (r-TMS) is a technique that allows non-invasive and relatively painless stimulation of cerebral cortex. It can reduce the experience of chronic pain by using magnetic field to produce small electrical currents in the cortex.The aim of this study is to determine the effectiveness of r-TMS treatment on patients with FBSS.

DETAILED DESCRIPTION:
Methods: In this double-blinded, randomized, placebo-controlled trial, 20 patients (aged 34-65 years) clinically diagnosed as FBSS, who had a history of surgery for LDH with persistent back and leg pain. Patients in r-TMS group received 5 Hz of r-TMS, as a 20-min (1000 pulses) daily session, 5 days per weeks, for a total of 10 sessions. R-TMS applied with MagVenture device (MagPro X100, Denmark, 2009) and figure eight coil (MMC 140 parabolic, MagVenture). Control group received sham r-TMS with the same protocol. Patients were assessed at baseline,after 5th and 10th sessions and 1 and 3 months after treatment. Visual Analogue Scale (VAS), DN-4 (Douleur Neuropathique-4 Questionnaire), Oswestry Disability Index (ODI), Beck Depression Inventory (BDI), Pittsburgh Sleep Quality Index (PSQI) were used for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 34-65 years
* Clinically diagnosed as FBSS
* History of surgery for LDH with persistent back and leg pain
* Patients with no root compression in postoperative magnetic resonance imaging of lumbar spine

Exclusion Criteria:

* Epilepsy
* Stroke
* Head trauma
* History of intracranial operation
* Cardiac pacemaker
* Pregnancy
* Postoperative lumbar root compression
* Neurologic deficits
* Prior physiotherapy for low back pain last 6 month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 months
  All groups were evaluated for low back and leg pain with Visual Analogue Scale (VAS) for rest, activity, and sleep-disturbing. Patients were instructed to indicate the severity of pain on a 10- point scale, on which 0 meant no pain, 5 meant moderate pain, and 10 meant intolerable pain.
Oswestry Disability Index | 4 months
  Functional status in all groups was evaluated with the Oswestry disability index (ODI). The ODI consists of 10 topics concerning pain, lifting, ability of selfcare, ability to walk, sit, stand and travel, social life, and sleep quality and is intended to assess disability and quality of life related to low back pain. ODI scores range from 0 (no disability) to 100 (maximum disability possible).
DN-4 Interview Questionnaire | 4 months
  The DN4-interview questionnaire (0-10) was used to identify neuropathic pain.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index | 4 months
  To evaluate the subjective amount of sleep, we used The Pittsburgh Sleep Quality Index (PSQI). The PSQI evaluates the sleep quality of the previous month, and it is clinically useful in the evaluation of several sleep disorders that affect sleep quality. It includes 19 self-administered questions and 5 questions to be answered by bedroom companions.
Beck Depression Inventory | 4 months
  Symptoms of depression were evaluated by means of the Beck Depression Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Yılmaz Kaysın, MD, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No
Patients in r-TMS group received 5 Hz of r-TMS, as a 20-min (1000 pulses) daily session, 5 days per weeks, for a total of 10 sessions. R-TMS was applied with MagVenture device (MagPro X100, Denmark, 2009) and figure eight coil (MMC 140 parabolic, MagVenture). Control group received sham r-TMS with the same protocol. Lumbar isometric exercises were given to all patients in both groups. Outcome measures were visual analogue scale (VAS) for rest, activity, and sleep-disturbing; Oswestry disability index; DN4-interview questionnaire; Pittsburgh Sleep Quality Index; Beck Depression Inventory (BDI).
  All patients were assessed at baseline, 5th session, 10th session, 1st and 3rd months after session.